CLINICAL TRIAL: NCT03072199
Title: Rituximab in Patients With Acute ST-elevation Myocardial Infarction Study
Acronym: RITA-MI
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Papworth Hospital NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P02100
Record Dates: First submitted 2017-02-24; First posted 2017-03-07 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Ischemic Heart Disease; Myocardial Infarction; Inflammation
Keywords: Rituximab; B cells
MeSH Terms: conditions — Myocardial Ischemia; Myocardial Infarction; Inflammation | interventions — Rituximab

STUDY DESIGN:
Intervention Model Description: Phase 1/2 unblinded interventional dose escalation study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Rituximab (Experimental)
  Interventions: Drug: RiTUXimab Injection

INTERVENTIONS:
Drug: RiTUXimab Injection — Single dose of Rituximab given intravenously within 48hours of myocardial infarction

SUMMARY:
RITA-MI aims to develop of a novel therapeutic concept to target the immune response in patients with acute myocardial infarction (MI) by depleting B-cells with a single injection of Rituximab which is approved for clinical use in cancer, autoimmune disease and inflammatory conditions. The goal is to re-purpose the drug, and translate the discovery into benefit for patients at high risk of cardiovascular events. Rituximab is expected to limit infarction size and improve the healing process, as complementary to other therapeutic strategies.

The applicants intend to perform a clinical study in patients with acute myocardial infarction (MI). The objective is to find the optimal dose (lowest dose with highest biological efficacy and best safety profile) for peripheral blood B cell depletion during the first 6 days after injection, and selective molecular signatures associated with improved heart function through analysis of peripheral blood samples.

The study rationale is to decrease the inflammatory reaction upon tissue necrosis following heart muscle ischemia.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years old
* Acute anterior (left anterior descending artery) STEMI and successful primary percutaneous coronary intervention (PCI) with stent implantation in the culprit lesion during the first 24h after onset of symptoms

Exclusion Criteria:

* A previous history of STEMI
* Cardiogenic shock (systolic blood pressure <80 mm Hg, unresponsive to fluids, or necessitating catecholamines), electrical instability or severe congestive heart failure
* Residual severe proximal bystander disease awaiting inpatient revascularisation
* Corrected QT interval (QTc) > 500 msecs using Bazett's formula
* Hematologic abnormalities (hemoglobin <10 g/dL or hematocrit <30%, platelet cell count of <100 x103/μL, white blood cell count <4 x103/μL)
* Hypogammaglobulinaemia (defined as <3g/L of IgG)
* Renal failure (estimated GFR by the MDRD formula < 45 ml/min/1.73m2);
* Known hepatic failure or abnormal liver function tests at baseline (ALT > 2 x ULN).
* Active or recurrent hepatitis (type B).
* Known HIV infection
* Current or previous tuberculosis (Chest X-Ray)
* Current infections
* Presence or history in the previous five years of an ongoing cancer, except in situ cancer of the cervix or basal cell carcinoma
* Any oral or intravenous immunosuppressive treatment (other than concomitant 100 mg methylprednisolone), disease modifying drugs, or other immune modulatory monoclonal antibodies or immunodepleting therapy at any time
* Allergy to rituximab or one of its excipients
* Expected need for vaccination with a live attenuated vaccine during the study including incomplete vaccination courses.
* Known or suspected pregnancy at screening or lactating woman
* Women of childbearing age unless confirmed by direct questioning that they are reproductively sterile or post-menopausal
* Participation in other clinical trials
* Inability to comply with study procedures

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Safety - Review of Adverse Events and Serious Adverse Events; | 6month
  Adverse and serious adverse events will be reviewed by daily history taking and clinical examination of patients whilst they are an inpatient. Subsequently patients will be followed up on discharge daily until day 6 with telephone follow up. On days 6, 14 and 6month patients will be assess again in an outpatient setting where adverse events will be documented. There is additional follow telephone follow up at day 30. After each group of 6 patients are recruited and infused with rituximab, an independent Data and Safety Monitoring Board will review the clinical and biological data and their side effect profile, including adverse events.
Safety - Clinically significant changes in biochemical and haematological markers | 6month
  Biochemistry and haematology bloods will be taken daily after drug administration whilst an inpatient. Upon discharge bloods will be taken on days 6, 14 and 6month for further assessment. Any new abnormalities will be flagged. After each group of 6 patients are recruited and infused with rituximab, an independent Data and Safety Monitoring Board will review the clinical and biological data and their side effect profile, including adverse events.
Safety - Clinically significant ECG changes | 6month
  Arrhythmia will be assess as patients will have continued cardiac monitoring whilst an inpatient. ECGs will be performed daily whilst an inpatient and also during outpatient attendance. QTc will be assessed using the Bazett formula. After each group of 6 patients are recruited and infused with rituximab, an independent Data and Safety Monitoring Board will review the clinical and biological data and their side effect profile, including adverse events.

SECONDARY OUTCOMES:
B cells | Days 0, 6, 14 and 6months
  Circulating B cells count before, immediately after administration (30 mins and 6 hours), and extended follow up (6 days, 14 days and 6months)
Cardiac biomarkers - Circulating inflammatory (hsCRP and IL6) and cardiovascular (BNP and Troponin) biomarkers. | Days 0, 2 and 6 months
  These will be measure before the infusion and compared to after infusion on days 2, 6 and 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Papworth Hospital NHS Trust, Cambridge, Cambridgeshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhao TX, Aetesam-Ur-Rahman M, Sage AP, Victor S, Kurian R, Fielding S, Ait-Oufella H, Chiu YD, Binder CJ, Mckie M, Hoole SP, Mallat Z. Rituximab in patients with acute ST-elevation myocardial infarction: an experimental medicine safety study. Cardiovasc Res. 2022 Feb 21;118(3):872-882. doi: 10.1093/cvr/cvab113. PMID 33783498